CLINICAL TRIAL: NCT06742151
Title: Evaluation of the Prevalence Rate and Related Risk Factors of Ridge Preservation
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, CHUNJUNG CHEN, Director of Periodontics, Chimei Medical Center
Other Study IDs: 1 0 3 0 3 - 0 0 5
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Dental Implants
Keywords: alveolar ridge preservation; Early implant placement
MeSH Terms: interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patient who received an implant after surgery.
  Interventions: Procedure: implant can be placed or not
- Group 2: Patient who didn't receive an implant due to insufficient bone volume or implant primary stability for implant placement.
  Interventions: Procedure: implant can be placed or not

INTERVENTIONS:
Procedure: implant can be placed or not — the possibility of receiving dental implants

SUMMARY:
Treated by dental implant is a well document and popular therapy nowadays. Placement of a dental implant in an ideal three-dimensional position is critical in achieving a predictable long-term success. However, healing of an extraction socket involves bone remodeling, which inevitably leads to atrophic changes of the alveolar ridge. Studies have shown that most of the resorption occurs during the first 3 months of healing, although dimensional changes can be observed up to 1 year after tooth extraction, resulting in approximately 50% reduction of the bucco-lingual dimension of the alveolar ridge, mainly due to the resorption of the bundle bone plate.

Therefore, the timing of implant placement in extraction sockets can influence the surgery operability and treatment period of time. The classifications of timing of implant placement in extraction sockets as following: Type I: immediate implant placement: implant placement immediately following tooth extraction and as part of the same surgical procedure. Type II: early implant placement: surgery after complete soft tissue coverage of the socket (typically 4~8 weeks).

Type III: early implant placement: implant surgery after substantial clinical and/or radiographic bone fill of the socket (typically 12~16 weeks). Type IV: late implant placement: surgery at healed site (typically more than 16 weeks). Considering of technique sensitivity and treatment time consuming, early implant placement is the most acceptable clinically.

Many techniques have been developed to maintain the architecture of residual alveolar ridges and regenerative techniques for socket preservation is one of them. This procedure has been widely tested in controlled and uncontrolled studies with various materials and clinical approaches. However, this procedure may require longer treatment period compare to conventional or early implant placement protocol. Meanwhile, there is no study revealed how often and when does socket preservation need to prevent the residual ridge deformity in our daily clinical practice. The aim of the study is try to retrospectively find out the possible advantages and percentage of ridge preservation after tooth extraction in order to understand whether the socket preservation technique is necessary after tooth extraction, and the possible factors which might affect the clinical decision-making.

DETAILED DESCRIPTION:
Background:

The alveolar process is a tooth-dependent tissue that develops in conjunction with the eruption of the teeth. The tooth is anchored to the jaws via the bundle bone into which the periodontal ligament fibers invest. Subsequent to the removal of the tooth, the alveolar process will undergo atrophy. The dynamics and magnitude of these changes have been investigated in the dog model as well as in humans. Most of the resorption occurs during the first 3 months of healing, although dimensional changes can be observed up to 1 year after tooth extraction, resulting in approximately 50% reduction of the bucco-lingual dimension of the alveolar ridge, mainly due to the resorption of the bundle bone plate. Some studies showed that significant loss of tissue contour occurs during the first month after tooth extraction, averaging 3~5mm in width at 6 months. As a result, a residual ridge is often inadequate for ideal implant placement, which creating a clinical challenge for the placement of a dental implant in an ideal position. However, placement of a dental implant in an ideal three-dimensional position is critical in achieving a predictable functional and esthetic restoration.

Therefore, the timing of implant placement in extraction sockets can influence the surgery operability and treatment period of time. The classifications of timing of implant placement in extraction sockets as following: Type I: immediate implant placement: implant placement immediately following tooth extraction and as part of the same surgical procedure. Type II: early implant placement: surgery after complete soft tissue coverage of the socket (typically 4~8 weeks).Type III: early implant placement: implant surgery after substantial clinical and/or radiographic bone fill of the socket (typically 12~16 weeks). Type IV: late implant placement: surgery at healed site (typically more than 16 weeks). Considering of technique sensitivity and treatment time consuming, early implant placement is the most acceptable clinically. However, different treatment strategies may be applied because of the vary amounts of resorption after tooth extraction.

Some of the extraction sockets will heal completely and the implant can be placed in an ideal position 3 months after tooth extraction. Others may require adjunctive surgical procedures (like guided bone regeneration, GBR) during the implant surgery. In some cases, with severe bone resorption after tooth extraction, staged approach for implant placement is recommended due to lack of sufficient bone volume, which is the most time consuming and expensive treatment method.

In order to avoid this situation, some surgical procedures have been described to prevent alveolar ridge collapsing after tooth extraction, including regenerative techniques for socket preservation and immediate implant placement after tooth extraction. The socket preservation technique has been widely tested in controlled and uncontrolled studies with various materials and clinical approaches. However, this may require longer treatment period compare to early implant placement protocol and so far, there is no study revealed how often and when does socket preservation need to prevent the residual ridge deformity in our daily clinical practice.

Purpose:

The purpose of this study is to evaluate:

1. How often do the clinical cases require ridge preservation than early implant placement protocol?
2. Which factors may influence the clinical decision?

Hypothesis:

Ridge preservation is better than early implant placement protocol.

Importance:

Help the clinician to make a more precise decision-making.

ELIGIBILITY:
Inclusion Criteria:

* periapical film at the time of tooth extraction
* implant surgery was scheduled within 4 months after tooth extraction.

Exclusion Criteria:

- who cannot identify the reason for tooth extraction or unclear periapical film

Ages: 21 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who plan to have single implant surgery from July 2009 to August 2015 were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
reason for tooth extraction | at the day of implant surgery
  due to caries, periodontal disease, tooth fracture, residual root, endodontic failure

SECONDARY OUTCOMES:
Radiographic analysis | at the day of implant surgery
  with or without apical lesion and with or without marginal bone loss

CONTACTS AND LOCATIONS:
Overall Officials: CHUNJUNG CHEN, MS, Principal Investigator — Chimei Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn JJ, Shin HI. Bone tissue formation in extraction sockets from sites with advanced periodontal disease: a histomorphometric study in humans. Int J Oral Maxillofac Implants. 2008 Nov-Dec;23(6):1133-8. PMID 19216285
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Buser D, Chappuis V, Belser UC, Chen S. Implant placement post extraction in esthetic single tooth sites: when immediate, when early, when late? Periodontol 2000. 2017 Feb;73(1):84-102. doi: 10.1111/prd.12170. PMID 28000278
- [Background] Cardaropoli G, Araujo M, Hayacibara R, Sukekava F, Lindhe J. Healing of extraction sockets and surgically produced - augmented and non-augmented - defects in the alveolar ridge. An experimental study in the dog. J Clin Periodontol. 2005 May;32(5):435-40. doi: 10.1111/j.1600-051X.2005.00692.x. PMID 15842256
- [Background] Cardaropoli G, Araujo M, Lindhe J. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 2003 Sep;30(9):809-18. doi: 10.1034/j.1600-051x.2003.00366.x. PMID 12956657
- [Background] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307